CLINICAL TRIAL: NCT01847924
Title: NEURoaid II (MLC 901) Assessment in Cognitively Impaired Not Demented Subjects : a Pilot Double Blind, Placebo-controlled Randomized Trial on Efficacy and Safety (NEURITES) Study
Brief Title: NEURoaid II (MLC 901) Assessment in Cognitively Impaired Not Demented Subjects
Acronym: NEURITES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MLC901-1
Record Dates: First submitted 2013-05-03; First posted 2013-05-07 (Estimated); Last update posted 2018-07-27 (Actual); Status verified 2018-06

CONDITIONS: Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Neuroaid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MLC901 (Active Comparator): Brand: Neuroaid II. Dosage: 2 capsules 3 times a a day
  Interventions: Drug: MLC901
- placebo (Placebo Comparator): MLC901 matching placebo made by the same manufacturer for this study dosage: 2 capsules 3 times a day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MLC901 — 24 weeks intervention with orally MLC901. 2 capsules 3 times a day
  Other Names: NeuroaidII (MLC901)
  Arms: MLC901
Drug: Placebo — 24 weeks intervention with orally placebo. 2 capsules 3 times a day
  Other Names: MLC901 matched Placebo
  Arms: placebo

SUMMARY:
Patients who have suffered from stroke may develop problems with thinking. Moreover, such patients have a high risk of becoming demented, more dependent or dying. Therefore, further studies are urgently needed to find effective and safe treatments.

Neuroaid is a Traditional Chinese Medicine which has been shown to stimulate growth of brain cells and connections in animals. Neuroaid may improve blood flow in the brain and functional recovery after stroke in patients. Neuroaid-II is a simplified formula with only the main 9 herbal ingredients of the original formula and no animal ingredients.

The NEURoaid II (MLC 901) assessment in cognitively Impaired not demented subjects: a pilot double blind, placebo-controlled randomized Trial on Efficacy and Safety (NEURITES) Study is a 24-week, early phase trial of Neuroaid-II in patients who have thinking problems after stroke. The study aims to investigate the effectiveness of the study drug in improving cognitive performance. The safety of the study drug will be closely monitored using adverse events, laboratory tests and vital signs.

The trial is important as it aims to set new standards for the scientific evaluation of Asian Traditional Medicine for integration into standard medicine practice. It may potentially establish a novel therapeutic approach for improving cognition after stroke.

DETAILED DESCRIPTION:
A substantial proportion of patients after non-disabling stroke are cognitively impaired compared to aged and education matched community dwelling controls. Moreover, post-stroke patients who have vascular cognitive impairment not dementia (VCIND) of moderate severity have a high risk of incident dementia, dependency and death. Further studies are urgently needed to demonstrate effective cognition enhancing therapies in VCIND given the absence of evidence based treatment options.

Neuroaid is a Traditional Chinese Medicine which has been shown to induce neurogenesis, promote cell proliferation and stimulate development of axonal and dendritic networks in animal models. Neuroaid may improve functional recovery after stroke in patients. Neuroaid-II is a simplified formulation with only 9 herbal and no animal ingredients.

The NEURoaid II (MLC 901) assessment in cognitively Impaired not demented subjects: a pilot double blind, placebo-controlled randomized Trial on Efficacy and Safety (NEURITES) Study is a 24-week Phase II study. The primary outcome is executive function as measured by the Verbal Fluency test. Secondary outcomes include cognitive measures such as the ADAS-Cog, MoCA, MMSE and a Cognitive Battery; Activities of Daily Living as measured by the ADCS-ADL scale; behaviour as measured by the Neuropsychiatric Inventory and depression as measured by the Geriatric Depression Scale and Beck Depression Scale. Safety and tolerability will be assessed using adverse events, laboratory tests, and vital signs.

The trial is important for translational medicine in Singapore through setting new standards for systematic evaluation of Traditional Medicine for integration into standard medicine practice

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients
2. Aged 55 to 85, living with a caregiver,
3. Modified Rankin score <=3.
4. Diagnosis of CIND due to cerebrovascular disease.
5. Cognitive impairment documented by neuropsychological evaluation within 12 months of index stroke/TIA. Not demented by DSM-IV criteria
6. Written informed consent by subject

Exclusion Criteria:

1. Advanced, severe, and unstable disease of any type that may interfere with the efficacy evaluations or put the subject at special risk.
2. DSM IV current diagnosis of dementia or major depression (patients may be included if currently being treated on an antidepressant and stabilized after 3 months).
3. A disability that may prevent the subject from completing all study requirements (e.g. blindness, deafness, severe language difficulty).
4. Ingestion of any of the following : an investigational drug in the past four weeks, a drug or treatment known to cause major organ system toxicity during the past four weeks, acetylcholinesterase inhibitors or memantine in the past 3 months

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Comparative change on executive function | Baseline to 24th week(24 week)
  To evaluate the comparative change from baseline with MLC901 and placebo on executive function in patients with cognitive impairment not dementia due to cerebrovascular disease, as measured by:
  Verbal Fluency and Colour Trails Test 1 & 2

SECONDARY OUTCOMES:
Comparative change on cognitive function | Baseline to 24th week(24 week)
  To evaluate the comparative change from baseline with Neuroaid and placebo on cognitive function, as measured by:
  ADAS-Cog MoCA Cognitive Battery (Symbol Digits Modalities Test, Maze, Digit Cancellation Test, Clock Drawing Test, Visual Memory Test and Frontal Assessment Battery)
Effects on activities of daily living | Baseline to 24th week(24 week)
  To evaluate the effects of Neuroaid on activities of daily living by :
  Alzheimer's Disease Cooperative Study Activities of Daily Living (ADCS-ADL) scale for mild cognitive impairment (MCI)
Effects on behaviour | Baseline to 24th week(24 week)
  To evaluate the effects of Neuroaid on behaviour by : Neuropsychiatric Inventory (NPI)
Effects on depression | 24 week
  To evaluate the effects of Neuroaid on depression by : Geriatric Depression Scale (GDS)
Adverse events, laboratory tests, and vital signs. | Baseline to 24th week(24 week)
  To evaluate the safety and tolerability of ML901 for 24 weeks of treatment, in comparison with placebo. Safety will be assessed using adverse events, laboratory tests, and vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher LH Chen, FRCP, Principal Investigator — National University Hospital, Singapore
Locations (5):
- University of Santo Tomas Hospital, Manila, National Capital Region, Philippines
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - National Neuroscience Institute, Singapore
- National Geriatric Hospital, Hanoi, Vietnam